CLINICAL TRIAL: NCT06128590
Title: Photobiomodulation for Controlling Pre-Local Anesthetic Injection Pain: A Double-Blind, Randomized Controlled Clinical Study
Brief Title: Photobiomodulation for Controlling Pre-Local Anesthetic Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5.598.425
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Fear Needles
Keywords: photobiomodulation, local anesthesics
MeSH Terms: conditions — Iatrophobia | interventions — Low-Level Light Therapy; Mepivacaine; Epinephrine; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: To randomly allocate participants into the experimental groups, a draw was conducted with 50 numbers using the Sealed Envelope website: https://www.sealedenvelope.com. The distribution was identical (1:1) for both groups, using a blocked design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The researcher responsible for administering FBM will be aware of the assigned interventions for each participant. Participants will remain unaware of the specific treatment they receive, as the treatment is standardized across both groups, with FBM being simulated in the control group. The outcome assessor will also be blinded to the interventions. Group identifications will be revealed only after the statistical analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Photobiomodulation (Group A) (Experimental): Participants will receive photobiomodulation therapy immediately before local anesthesia, in the same place where the puncture will be performed for pterygomandibular anesthesia.
  Interventions: Device: Photobiomodulation; Drug: Mepivacaine hydrochloride in combination with epinephrine
- Control: Laser Sham (Group B) (Sham Comparator): The participants will be treated in the same way as in group A. The person responsible for applying the PBM will simulate the irradiations by positioning the device in the same place as described for the experimental group, but the equipment will be switched off. So that the participant does not identify the group to which they belong, the device's activation sound (beep) will be simulated by the device itself, which makes the beep sound by pressing the activation button only once. After this, pterygomandibular anesthesia will be carried out in the same way.
  Interventions: Drug: Mepivacaine hydrochloride in combination with epinephrine; Device: Photobiomodulation simulation

INTERVENTIONS:
Device: Photobiomodulation — Photobiomodulation was applied before the procedures at an infrared wavelength of 808nm, at a power of 100mW, 1 point with a total energy of 8J, time of 80s, irradiance of 3.33W/cm² and radiant exposure of 266.66 J/cm2. The application point was on the retromolar region where the needle was inserted to perform the anesthetic, in a single application before the procedure.
  The patient and operator were properly protected with goggles in both the control and experimental groups.
  Arms: Experimental: Photobiomodulation (Group A)
Drug: Mepivacaine hydrochloride in combination with epinephrine — The anesthetic of choice will be Mepivacaine, which is widely used in dentistry with duration between 1.5 and 2 minutes. The maximum recommended dose is 6.6 mg/Kg, not exceeding 400 mg or 11 anesthetic tubes.
  It is a sterile injectable solution of 2% mepivacaine hydrochloride (20 mg/mL) in combination with epinephrine 1:100,000 (0.01 mg/mL). Each vial contains 1.8 mL, 36 mg of mepivacaine hydrochloride, and 0.018 mg of epinephrine. All patients will use anesthetics from the same brand (DLA Pharmaceutical LTDA), one of the most widely used on the market. All patients will be anesthetized with tubes from the same batch, one tube per procedure.
  Other Names: Local anesthetic
Device: Photobiomodulation simulation — The participants will be treated in the same manner as in group A. The person responsible for the application of FBM will simulate the irradiations by placing the device in the same location described for the experimental group, but the equipment will remain turned off. To prevent the participant from identifying their group, the activation sounds of the devices (beeps) will be recorded to simulate the device's operation.
  Arms: Control: Laser Sham (Group B)

SUMMARY:
The objective of this study is to assess whether pre-anesthetic photobiomodulation (PBM) can effectively reduce needle puncture pain and enhance the efficiency of local anesthesia. In this double-blind randomized controlled trial, 50 participants were included. The control group underwent the standard anesthetic procedure, while the experimental group received the application of an infrared laser (100mW at 808nm, 8J at a single point) immediately before anesthesia, at the site of the intended needle puncture. Both groups underwent the same anesthetic procedure, administered by the same operator. The outcome evaluator and the patient were blind to the FBM application. The primary outcome of the study focused on pain experienced at the time of needle insertion, assessed using the Visual Analogue Scale (VAS) during the needle's introduction. Secondary outcomes encompassed anxiety levels, measured using the Beck questionnaire, anesthetic onset time determined through the electric pulp test, the number of anesthetics required for the procedure, and the necessity for supplementary anesthesia.

DETAILED DESCRIPTION:
Dental fear and phobia are widespread worldwide, with local anesthesia being one of the procedures that patients fear the most. To alleviate the pain associated with needle insertion and the need for repeat procedures, various complementary therapies have been introduced. However, to date, there is no established protocol for this intervention. The objective of this study is to assess whether pre-anesthetic photobiomodulation (PBM) can effectively reduce needle puncture pain and enhance the efficiency of local anesthesia. In this double-blind randomized controlled trial, 50 participants were included. The control group underwent the standard anesthetic procedure, while the experimental group received the application of an infrared laser (100mW at 808nm, 8J at a single point) immediately before anesthesia, at the site of the intended needle puncture. Both groups underwent the same anesthetic procedure, administered by the same operator. The outcome evaluator and the patient were blind to the FBM application. The primary outcome of the study focused on pain experienced at the time of needle insertion, assessed using the Visual Analogue Scale (VAS) during the needle's introduction. Secondary outcomes encompassed anxiety levels, measured using the Beck questionnaire, anesthetic onset time determined through the electric pulp test, the number of anesthetics required for the procedure, and the necessity for supplementary anesthesia. Categorical variables will be presented as absolute and relative frequencies and compared using the Pearson chi-squared test, likelihood ratio test, or Fisher's exact test. Quantitative variables will be assessed for normality using the Kolmogorov-Smirnov test. Outcome variables will be presented as mean and standard deviation or median and interquartile range (IQR) and compared using the Student's t-test or Mann-Whitney test. Variables measured under multiple conditions will be compared using analysis of variance for repeated measures. A significance level of P < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 60 years old
* Both genders
* Without comorbidities
* Who required pterygomandibular anaesthesia for a dental procedure.

Exclusion Criteria:

* Any sign of pain or inflammation at the puncture site (e.g. presence of pericoronaritis)
* Active periodontitis/gingivitis
* Use of a pacemaker
* Use of prostheses, fixed metal appliances
* Using anti-inflammatory, analgesic or corticosteroid therapy for less than 1 week.
* Pregnant and/or breastfeeding women
* Need to use a local anaesthetic other than Mepivacaine with vasoconstrictor (anaesthetic of choice for the study)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Immediately Before anesthesia
  It will be carried out as follows: the healthcare professional asks the patient to select a point on a line 10cm long, drawn between two extremities to express the intensity of the pain. Patients will be asked to rate "current" pain intensity or, in other cases, pain intensity "in the last 24 hours". The VAS is a simple-to-use assessment tool that does not require sophisticated equipment. It is also highly sensitive in detecting the effects of treatment, and its results can be analyzed using parametric tests. In this study, a plastic band was made for all patients,
Pain assessment | Immediately After anesthesia
  It will be carried out as follows: the healthcare professional asks the patient to select a point on a line 10cm long, drawn between two extremities to express the intensity of the pain. Patients will be asked to rate "current" pain intensity or, in other cases, pain intensity "in the last 24 hours". The VAS is a simple-to-use assessment tool that does not require sophisticated equipment. It is also highly sensitive in detecting the effects of treatment, and its results can be analyzed using parametric tests. In this study, a plastic band was made for all patients,

SECONDARY OUTCOMES:
Anxiety assessment using Beck's questionnaire | Immediately Before anesthesia
  Anxiety analyses will be carried out using the BAI (by Beck, Epstein, Brown & Steer, 1988), adapted and validated for Brazil by Cunha (2001), which will be applied before and after treatment.
  The BAI is a multiple-choice questionnaire containing 21 questions about common anxiety symptoms. The score ranges from 0 to 63, and is classified as minimal anxiety (score: 0-10), mild anxiety (score: 11-20), moderate anxiety (score: 21-30) and severe anxiety (score: 31-63). The questionnaire will be answered by the participants themselves, who will read the questions and answer them manually before starting the research and after the end of the treatment. At the end of the treatment, the score obtained will be calculated and applied to the results collection form.
Anxiety assessment using Beck's questionnaire | Immediately After anesthesia
  Anxiety analyses will be carried out using the BAI (by Beck, Epstein, Brown & Steer, 1988), adapted and validated for Brazil by Cunha (2001), which will be applied before and after treatment.
  The BAI is a multiple-choice questionnaire containing 21 questions about common anxiety symptoms. The score ranges from 0 to 63, and is classified as minimal anxiety (score: 0-10), mild anxiety (score: 11-20), moderate anxiety (score: 21-30) and severe anxiety (score: 31-63). The questionnaire will be answered by the participants themselves, who will read the questions and answer them manually before starting the research and after the end of the treatment. At the end of the treatment, the score obtained will be calculated and applied to the results collection form.
Latency time | Immediately Before anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Latency time | 2 minutes after anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Latency time | 5 minutes after anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Latency time | 10 minutes after anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Latency time | 15 minutes after anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Latency time | 20 minutes after anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Latency time | 25 minutes after anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Latency time | 30 minutes after anesthesia
  To establish a standard, the tests will be carried out on permanent premolars, with normal reaction scales ranging from 20 to 50. For convenience in terms of ease of visualization, the first lower premolar was preferably chosen; if the element was absent, it was carried out on the second lower premolar. Data was collected before treatment and at 2, 5, 10, 15, 20, 25 and 30 minutes after anaesthesia, timed using a digital stopwatch on a mobile phone.
  The thermal test will be carried out before the procedure to double-check the pulp vitality of the elements, as stated in the literature.The cold test will be carried out with cotton wool on the buccal surface of the first premolar or the same as the electrical test, for 15 seconds or until the patient indicates that they feel sensitivity.
Assessment of blood pressure | Immediately Before anesthesia
  A manual sphygmomanometer was used, and assessed by the same professional.
Assessment of blood pressure | 10 minutes after anesthesia
  A manual sphygmomanometer was used, and assessed by the same professional.
Blood oxygen saturation level | Immediately Before anesthesia
  For this purpose, digital oximeter were used, and assessed by the same professional.
Blood oxygen saturation level | 10 minutes after anesthesia
  For this purpose, digital oximeter were used, and assessed by the same professional.
Pterygomandibular technique success rate | Immediately After procedure
  The anesthetic success rate will be calculated by counting the number of times the procedure has been effective, i.e. if 30 minutes after anesthesia, the electrical test does not determine a mark of 50 on the display, this means that the anesthetic technique has failed. Even if the patient reports that the tissues are anesthetized, for complete pterygomandibular anesthesia, it is necessary to anesthetize the pulp, the lingual region, the vestibular region and the corresponding lower lip. If there is no complete anesthesia, this patient will be considered a "failure of anesthesia", but the patient will not be excluded from the study, since the main outcome of pain has already been collected without interference.
Suplementar anesthesia | Immediately after procedure
  Number of anesthetic tubets needed for anesthetic supplementation during the procedure was counted

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina Horliana, PhD, Study Director — University of Nove de Julho
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil